CLINICAL TRIAL: NCT05205707
Title: Association of Circulating ACE2 Levels With COVID-19
Status: Completed | Type: Observational
Sponsor: Jordan University Hospital (Other)
Responsible Party: Principal Investigator, Amjad Banihani, Associate professor, Jordan University Hospital
Other Study IDs: 2021/5
Record Dates: First submitted 2022-01-22; First posted 2022-01-25 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; COVID-19 Respiratory Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 Patients: Blood sample from admitted patients will be drawn
  Interventions: Diagnostic Test: ACE serum levels
- Control Patients: Blood sample from control group will be drawn
  Interventions: Diagnostic Test: ACE serum levels

INTERVENTIONS:
Diagnostic Test: ACE serum levels — Circulating ACE2 level will be measured

SUMMARY:
COVID-19 cases are rising substantially in Jordan. Since this is a novel virus, there is still much to be investigated surrounding its pathophysiology in order to attempt to find suitable treatments or better decision-making in the prognosis of the disease. This project aims to identify if soluble angiotensin-converting enzyme (ACE2) can be used as a prognostic factor for COVID-19 severity, which will allow clinicians to manage COVID-19 cases more efficiently. ACE2 is of interest since the coronavirus enters host cells through ACE2 receptors. It can slo be hypothesized that the irus may also bind to soluble ACE2, but without mediating its effects. It si, therefore, expected that those with higher levels of ACE2 would more likely have milder disease. This can potentially help improve survival rate, allowing clinicians to identify the higher-risk patients and monitoring them more closely.

DETAILED DESCRIPTION:
SARS-CoV-2 is a new isolate of coronavirus that caused an epidemic in Wuhan, China in December 2019. The virus has then spread to the rest of the world causing a pandemic, and the disease the virus causes was designated the name COVID-19.

The presence of underlying medical condition increases a risk of severe disease course. Diabetes and cardiovascular disease are amongst the conditions that are associated with the worst COVID-19 prognosis . Renal failure is also associated with more severe illness On another note, angiotensin-converting enzyme 2 (ACE2) is expressed in human airway epithelia, lung parenchyma, small intestine cells as well as in the heart, kidneys and testis It functions as both an enzyme and a receptor for viral entry as it is known that SARS-CoV-2 enters into human host cells mainly through the cellular receptor ACE2, . It is hypothesized that with the damage and loss of cells induced by infection, enzymatic ACE2 activity would be globally compromised, inducing a state of relative ACE2 deficiency. This leads to enhanced and protracted tissue and vessel exposure to Ang II and therefore vasoconstriction, enhanced thrombosis, increased tissue permeability and cytokine production resulting in inflammation Chronic angiotensin 1 receptor (AT1R) blockade elevates ACE2 expression . Unlike ACE1, however, ACE2 is insensitive to the actions mediated by ACE inhibitors . It might be appealing to propose that chronic use of ACE inhibitors or AT1R antagonists puts patients at particular high risk if they get infected with SARS-CoV-2, as ACE2 overexpression may facilitate viral replication in the lung tissue . However, results of some studies performed in healthy human subjects did not confirm such results. In vitro studies, on the other hand, depict reduced concentrations of soluble ACE2 despite the increase in membrane expression and tissue levels. Therefore, there is no current significant evidence regarding the effects of ACE inhibitors and ARBs on COVID-19 infection .

In contrast, mild or moderate ACE2 deficiency is unlikely to be protective from viral invasion either. This is due to the intrinsically high affinity of SARS-CoV-2 to ACE2 receptors The soluble form of ACE2 may be a biomarker of severity of COVID-19 progression in patients . This could be due to the fact that COVID-19 binds to the soluble form, leaving less to be bound to the ACE2 receptor and be taken up by host cells The aim of this project is to identify any association between ACE2 levels with severity of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 and above
* Gender: both males and females.
* Confirmed diagnosis of COVID-19 for patients and confirmed absence of COVID-19

Exclusion Criteria:

* Healthy individuals: not being diagnosed with COVID-19 or at least has not been in close contact with a person diagnosed with COVID-19.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All adult COVID 19 patients admitted to Jordan University Hospital during 3 months.
Sampling Method: Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
ACE2 level | 3 months
  Serum level of ACE2 in control and COVID 19 patients will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Jordan, Amman, Jordan